CLINICAL TRIAL: NCT07215429
Title: SpO2 Validation Study - Philips Optimus
Brief Title: SpO2 Validation Study-Philips Optimus
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: Protocol # PR 2024-608_300178
Record Dates: First submitted 2025-09-08; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Pulse Oximetry, Oxygen Measurements, SpO2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Philips Wireless Patient Module SpO2 (Gen-4): This device is a complete pulse oximeter measurement module that utilizes the Philips PicoSAT II+ SpO2 processor that is a component on the circuit car assembly, part number 453665151651. This processor incorporates all signal processing and algorithms to derive the oxygen saturation value (SpO2), pulse rate, perfusion indicator value, and the plethysmographic waveform
  Interventions: Device: No intervention
- SpO2 Sensor, MRI (Gen-4): This is a fiber-optic cable that is attached via an connector at one end to the Philips Wireless SpO2 Patient Module, and one of the SpO2 finger accessories at the other end. This cable serves as the conduit through which red and infrared light is transmitted into the finger and then is received back from the other side of the finger into the photodiode. The red and infrared LEDs and the photodiode are all contained in the cable housing. The cable itself is made from RoHS-compliant fiber-optic materials. Fiber-optics are utilized to allow the SpO2 module to operate properly in the MRI environment.
  Interventions: Device: No intervention
- SpO2 Accessories: SpO2 Grips (Single Use) and SpO2 Gloves (Reusable): The SpO2 Grips and Gloves are designed to securely hold the SpO2 Sensor in proper location when it is attached to the Wireless SpO2 module. Both finger accessories provide two slide-in clip attachments for connecting to the SpO2 Cable ends, designed to be positioned at the top and bottom of the finger. The reusable finger accessory is designed to slide onto the finger and secure itself by means of a rubber-like material that provides the appropriate grip
  Interventions: Device: No intervention
- Silver Reference: IntelliVue Patient Monitor X3 and Adult SpO2 Sensor (M1191BL): The IntelliVue X3 is a versatile patient monitoring device with a color touchscreen display. It can simultaneously monitor ECG (using 3-, 5-, 6- or 10-lead sets, including arrhythmia and ST monitoring), respiration, SpO2, NBP, two invasive pressures, temperature, and CO2. The multi-touch screen allows easy interaction by swiping and tapping with one or two fingers.
  Interventions: Device: No intervention

INTERVENTIONS:
Device: No intervention — No intervention

SUMMARY:
Validation study to validate the SpO2 accuracy performance of the Sponsor's SpO2 sensors over the range of 70-100% SaO2 during non-motion conditions assessed by CO-Oximetry

DETAILED DESCRIPTION:
The intent of this clinical study is to validate the SpO2 accuracy performance of the Sponsor's SpO2 sensors over the range of 70-100% SaO2 during non-motion conditions assessed by CO-Oximetry. The end goal is to provide supporting documentation for the SpO2 accuracy validation of the Sponsor's pulse oximeter with consideration to anticipated updates to ISO 80601-2-61:2025(E)

ELIGIBILITY:
INCLUSION CRITERIA

Participants accepted in this study must meet all the following criteria:

* Participant must have the ability to understand and provide written informed consent.
* Participant is an adult between 18-50 years of age.
* Participant must be willing and able to comply with study procedures and duration.
* Participant is a non-smoker or who has not smoked within 2 days prior to the study.

EXCLUSION CRITERIA

* Participant is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation (i.e., Raynaud's Syndrome), injury, open wound, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. Tattoos in the optical path which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow participants to participate if the condition is noted and would not affect the sites utilized.)
* Females who are pregnant
* Females who are trying to get pregnant (with confirmation of positive urine pregnancy test unless the participant is known to be not of child-bearing potential)
* Participants who have smoked in the last 2 days or participants who have refrained, for at least 48 hours, with COHb levels >3% as assessed with a Masimo Radical 7 (Rainbow)
* Participants with known respiratory conditions such as: (self-reported)

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * unresolved respiratory or lung surgery,
  * emphysema, COPD, lung disease
  * Recent COVID with or without hospitalization (last 2 months)
* Participants with self-reported heart or cardiovascular conditions such as: (self-reported, except for blood pressure and ECG review)

  * high blood pressure: systolic >140 mmHg or diastolic >90 mmHg on 3 consecutive readings (reviewed during health screen)
  * have had cardiovascular surgery, except successful minor surgery without clinical symptoms (i.e., PFO, PDA)
  * chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia (reviewed during health screen)
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
  * implantable active medical device such as pacemaker or automatic defibrillator
* Self-reported health conditions as identified in the Health Assessment Form

  * diabetes,
  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent symptomatic head injury (within the last 2 months),
  * Cancer requiring chemotherapy, radiation, or current treatment.
* Participants with known clotting disorders (self-reported)

  * history of bleeding disorders or personal history of prolonged bleeding from injury
  * history of blood clots
  * hemophilia
  * current use of blood thinner: prescription or daily use of aspirin
  * Sickle Cell Trait or Disease
* Participants with severe contact allergies to standard adhesives, latex, silicone or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported)
* Participants with severe allergies to iodine (only applicable if iodine is used)
* Participants with severe allergies to lidocaine (or similar pharmacological agents, e.g. Novocaine),
* Failure of the Perfusion Index Ulnar/Ulnar+Radial Ratio test (Ratio <0.4)
* Unwillingness or inability to remove nail polish or artificial nails from test digits.
* Participant received intravascular dye within the past 48 hours (e.g. Indocyanine green, methylene blue, dyes used in cardiac output monitoring)
* Surgical hardware in pathway of Device Under Test
* Other known health conditions should be considered upon disclosure in health assessment form.
* Participants with uneven skin tone at the sensor site or at the forehead

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: minimum of 66 participants up to a maximum of 180, healthy male and female volunteers of any race, ranging in pigmentation from light to dark. he study population will meet the following stratification criteria:
  * At least 25% of the population with Monk 1-3 with ITA > 30 at the forehead
  * At least 25% of the population with Monk 4-7 with ITA ≤ 30 and ≥ -30 at the forehead
  * At least 25% of the population with Monk 8-10 with ITA < -30 at the forehead
    * At least half of the participants in this group will have an ITA < -50 at the forehead
    * In the event the Monk and ITA place a participant in different cohorts, the ITA shall be used to determine the demographic cohort for the participant
  * At least 40% of the population male
  * At least 40% of the population female
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2025-09-09 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
SpO2 accuracy of the SpO2 sensors under test with the Philips MRI Patient Monitoring | Day 1
  Pulse Oximetry Subsystem during non-motion conditions over the range of 70-100% SaO2, when compared with the reference SaO2 obtained from CO-Oximetry analysis of arterial blood samples.

SECONDARY OUTCOMES:
evaluate non-disparate performance (differential bias) of the SpO2 sensors under test | Day 1
  with the Philips MRI Patient Monitoring Pulse Oximetry Subsystem during non-motion conditions in the SaO2 ranges of 70% ≤ SaO2 ≤ 85% and 85% < SaO2 ≤100%.
  with the Philips MRI Patient Monitoring Pulse Oximetry Subsystem during non-motion conditions in the SaO2 ranges of 70% ≤ SaO2 ≤ 85% and 85% < SaO2 ≤100%.
  with the Philips MRI Patient Monitoring Pulse Oximetry Subsystem during non-motion conditions in the SaO2 ranges of 70% ≤ SaO2 ≤ 85% and 85% < SaO2 ≤100%.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Rabanal, NP, Principal Investigator — Element Desaturation Labratory
Locations (1):
- Element Materials Technology, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No